CLINICAL TRIAL: NCT02409771
Title: Prospective Multicenter Clinical Trial With the PRECIZON Presbyopic Multifocal Intraocular Lens
Brief Title: Clinical Trial With PRECIZON Presbyopic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ophtec BV (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AP01000538
Record Dates: First submitted 2015-03-12; First posted 2015-04-07 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-04

CONDITIONS: Cataract; Presbyopia
MeSH Terms: conditions — Cataract; Presbyopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention arm (Experimental): Bilateral implantation with PRECIZON Presbyopic intraocular lens
  Interventions: Device: PRECIZON Presbyopic

INTERVENTIONS:
Device: PRECIZON Presbyopic — Optical correction of aphakia in adults in whom the crystalline lens has been removed and who desire presbyopia correction.
  Other Names: PRECIZON Presbyopic Multifocal intraocular lens (MIOL)

SUMMARY:
The purpose of this clinical trial is to evaluate the effectiveness of the PRECIZON Presbyopic.

DETAILED DESCRIPTION:
Prospective, open-label, single-arm, multicenter clinical evaluation with a 3 months follow-up. The PRECIZON Presbyopic is a lens intended for implantation in the capsular bag, indicated for optical correction of aphakia in adults whom the crystalline lens has been removed and who desire presbyopia correction. The main objective is to evaluate the ability of the PRECIZON Presbyopic to provide near, intermediate and distance vision in patients undergoing cataract extraction / Clear Lens Exchange (CLE) and intraocular lens implantation. Study results will be used for CE-approval and registration and marketing purposes.

ELIGIBILITY:
Inclusion Criteria:

* Presbyopic
* Cataract patient or Clear Lens Extraction (CLE) candidate
* Patients wishes to be spectacle independent for near and far vision
* Patient lifestyle and outlook fit with multifocal IOL implantation
* Qualifies for bilateral implantation
* Patient must have a calculated IOL power within the available diopter range
* Expected best corrected visual acuity of 0.5 Snellen decimal or better after IOL implantation.
* No secondary surgical procedure planned during the course of the study
* Availability, willingness and sufficient cognitive awareness and physical ability to comply with examination procedures throughout the entire duration of the study
* Patients must provide written informed consent
* The predicted keratometric postoperative astigmatism (calculated with respect to the surgical induced astigmatism) must be <1.0 D.

Exclusion Criteria:

* Ocular disease other than cataract that may predispose for future complications or might confound the outcome of the investigation (e.g. anterior segment pathology, glaucoma, corneal dystrophy, ocular inflammation, pseudoexfoliation syndrome, retinal disorders)
* Acute or chronic disease or illness or use of medication that could confound the outcome of the study or increase the risk to the subject
* Endothelial cell count <1500 cells/mm2
* Amblyopia
* Congenital eye abnormalities
* Previous ocular surgery that might confound the outcome of the investigation or increase risk to patient
* Concurrent participation or participation during the last 30 days in any other clinical trial
* Patient must not be pregnant or has another condition with associated fluctuation of hormones that could lead to refractive changes

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2017-01-17 (Actual); Study Completion 2017-01-17 (Actual)

PRIMARY OUTCOMES:
Improvement in monocular and binocular uncorrected and corrected near visual acuity | 3 months follow-up postoperative
  The ability of the PRECIZON Presbyopia Intraocular lens (IOL) to provide near visual acuity
Improvement in monocular and binocular uncorrected and corrected intermediate visual acuity | 3 months post-op
  The ability of the PRECIZON Presbyopia Intraocular lens (IOL) to provide intermediate visual acuity
Improvement in monocular and binocular uncorrected and corrected distance visual acuity | 3 months post-op
  The ability of the PRECIZON Presbyopia Intraocular lens (IOL) to provide distance visual acuity

SECONDARY OUTCOMES:
Photopic contrast sensitivity as measured by a contrast sensitivity chart | 3 months postoperative
  Binocular contrast sensitivity scores for spatial frequencies of 3.0 cpd, 6.0 cpd, 12.0 cpd and 18.0 cpd.
Mesopic contrast sensitivity as measured by a contrast sensitivity chart | 3 months post-op
  Binocular contrast sensitivity scores for spatial frequencies of 3.0 cpd, 6.0 cpd, 12.0 cpd and 18.0 cpd.
Stability of manifest refraction (MRSE) as measured by a mean change in MRSE between visits as determined by a paired analysis | 3 months post-op
  Percentage of eyes that achieve a change of less than or equal to 1.00 D of MRSE between two refractions performed 3 months apart
Spectacle dependency | 3 months post-op
  Percentage of patients that achieve complete spectacle independence or occasional use of glasses for near or intermediate vision
Defocus curve | 3 months post-op
  Binocular defocus evaluation will be obtained by using the best corrected distance refraction and then defocusing the image in 0.5 D increments to -0.5 D.
Rates of adverse events and complications | 3 months post-op
Patient satisfaction as measured by a patient satisfaction questionnaire | 3 months post-op
Quality of vision as measured by the Quality of Vision (QoV) questionnaire | 3 months post-op
  Percentage of patients with a QoV score >10 and >30 at 3 months postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Mike P. Holzer, Prof. Dr., Principal Investigator — Heidelberg University
Locations (6):
- Medipolis, Wilrijk, Belgium
- Universitäts-Augenklinik Heidelberg, Heidelberg, Germany
- Academisch Ziekenhuis Maastricht, Maastricht, Limburg, Netherlands
- Spain (2):
  - Oftalvist CIO Jerez, Jerez de la Frontera
  - Hospital Universitari Mútua Terrassa, Terrassa
- Acibadem Maslak Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided